CLINICAL TRIAL: NCT05675982
Title: Real-Time Monitoring of Circulating Tumor DNA and Study of Prognostic Factors in Patients Treated With Anti-CD19 CAR-T Cells for Relapsed or Refractory Diffuse Large B-cell Lymphoma
Brief Title: Real-Time Monitoring of Circulating Tumor DNA and Study of Prognostic Factors in Patients Treated With CAR-T Cells
Acronym: RT-CAR
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Henri Becquerel (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CHB22.02
Record Dates: First submitted 2022-12-22; First posted 2023-01-09 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Diffuse Large B Cell Lymphoma
Keywords: Circulating tumor DNA; Diffuse Large B Cell Lymphoma; next generation sequencing; liquid biopsy
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Minimal residual disease assessment (Experimental)
  Interventions: Other: CAR-T cells monitoring

INTERVENTIONS:
Other: CAR-T cells monitoring — monitoring of circulating DNA by blood sample

SUMMARY:
The purpose of this study is to demonstrate that it is possible to report in real time (less than 3 weeks) to the hematologist the results of the molecular minimal residual disease (MRD) based on blood circulating tumor DNA (ctDNA) assessment taken approximately 7 days after the reinjection of the CAR-T cells, in order to be able to anticipate a possible progression of the disease and to be able to propose salvage or earlier adjuvant therapy to improve patient prognosis.

DETAILED DESCRIPTION:
The main objective is to demonstrate the feasibility of monitoring residual disease in real time by monitoring circulating tumor DNA in patients with relapsed or refractory diffuse large cell B-cell lymphoma treated with anti-CD19 CAR-T (axi-cel, tisa -cel or liso-cel).

The primary endpoint of the study is to assess the capacity of our research lab to transmit the result of the molecular characterization of the residual disease (MRD) sampled on Day+7 (+/- 3 days) of the injection of CAR-Ts (MRD evaluated by the quantity of ctDNA by NGS technique) of the patient with DLBCL R/R treated with CAR-T, to the recruiting investigator no later than Day+28 (+ /- 3 days). We will evaluate the proportion between the number of informative evaluable patients (patients with at least one detectable mutation in pre-treatment and having reached the PET-CT evaluation of Day+28) and the total number of informative patients (patients with at least one mutation detectable in pre-treatment). The target will be achieved and real-time MRD assessment will be considered feasible if the proportion is at least 80%.

Patients who do not have a detectable mutation in pre-treatment ("non-informative patients for follow-up of residual disease"), as well as patients who do not reach the ctDNA sample by Day+7, and/or do not not reaching the PET-CT by Day+28, will be considered as not evaluable for the primary endpoint, and will be the subject of a separate descriptive analysis and will be evaluable for the secondary objectives. We took this into account when evaluating the number of patients to include.

Day0 corresponds to the day of injection of the CAR-Ts, Day+7 corresponds to the 8th day post-injection of the CAR-Ts, and D+28 refers to the planned date of the PET-CT evaluation of Day+28 (this examination being the "gold standard" for the evaluation of the response to treatment with CAR-T).

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 or over
* Carriers of relapsed or refractory diffuse large cell B-cell lymphoma (LBDGC R/R), relapsed or refractory primary mediastinum B-cell lymphoma or follicular lymphoma transformed into LBDGC R/R
* Patients with an indication for treatment with CAR-T anti CD19
* PET-CT pre-injection of CAR-T performed
* Signed informed consent
* Patients affiliated or beneficiaries of a health insurance scheme

Exclusion Criteria:

* Pregnant or breastfeeding women
* Absence or insufficiency of tumor material (patient's most recent diagnostic biopsy) fixed in FFPE paraffin of insufficient quality/quantity for next-generation sequencing (NGS) analysis
* Lack of patient consent
* Patient treated with CAR-T as part of a therapeutic clinical trial
* Patient whose weight is less than 30 kg
* Protected adult or deprived of liberty (under guardianship or curatorship)
* Patient unable to understand the study for any reason whatsoever or to comply with the constraints of the trial (language, psychological, geographic problem, etc.).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2023-01-13 (Actual); Primary Completion 2025-09-08 (Actual); Study Completion 2026-09-08 (Estimated)

PRIMARY OUTCOMES:
Time required to report minimal residual disease report | 28 days
  To to assess the capacity of the research lab to transmit the result of the molecular characterization of the residual disease sampled on day 7 of the injection of CAR-Ts of the patient to the recruiting investigator no later than day 28.

SECONDARY OUTCOMES:
Progression free survival | one year
  time between inclusion and progression
Overall survival | one year
  time between inclusion and death with all cause of mortality

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Camus, MD, Principal Investigator — Centre Henri Becquerel
Locations (1):
- Centre Henri Becquerel, Rouen, France

IPD SHARING:
Plan to Share IPD: No